CLINICAL TRIAL: NCT06160401
Title: Safety, Tolerability and Pharmacokinetic Characteristics of Singletine(DC407) in Healthy Adult Subjects After Single and Multiple Doses: a Single-center, Randomized, Double-blind, Placebo-controlled, Phase 1 Trial
Brief Title: Evaluation of Safety, Tolerability, PK/PD, and Metabolism of Single-Dose Singletine(DC407) in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JYC0101
Record Dates: First submitted 2023-11-04; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Singletine（DC407） ascending dose (Experimental): Single ascending dose
  Interventions: Drug: Singletine
- Singletine（DC407）food influence group (Experimental): Food influence group
  Interventions: Drug: Singletine
- Singletine placebo comparator(Single ascending dose) (Placebo Comparator): Single ascending dose
  Interventions: Drug: Placebo
- Singletine placebo comparator(food influence group) (Placebo Comparator): Food influence group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Singletine — Singletine orally administered
  Other Names: Singletine（DC407）experimental group
  Arms: Singletine（DC407） ascending dose; Singletine（DC407）food influence group
Drug: Placebo — Placebo orally administered
  Other Names: Placebo group
  Arms: Singletine placebo comparator(Single ascending dose); Singletine placebo comparator(food influence group)

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetic characteristics of Singletine in healthy adult subjects. The main questions it aims to answer are: safety and tolerability of Singletine in healthy subjects, the pharmacokinetic characteristics after single and multiple doses and the effect of food on the pharmacokinetic characteristics. Participants will be treated with Singletine orally and safety and pharmacokinetic evaluations will be conducted according to the protocol.

DETAILED DESCRIPTION:
This study will be an double-blinded, single-center phase I clinical trial. After being informed about the study and potential risks, all subjects giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry. And then subjects will be administered for single-dose treatment or 7-day multiple-dose treatment and 9-day safety follow up after the last dose of treatment. The safety and pharmacokinetic measures will be conducted according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old (including both endpoints), healthy males or females;
* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) between 19-28 kg/m2 (including both endpoints);
* No significant abnormal clinical symptoms, normal physical examination, vital signs, 12-lead electrocardiogram (ECG), chest CT, ultrasound, and important indicators in laboratory tests show no clinically significant abnormalities;
* Subjects (including partners) have no parenting plans within 90 days from screening to the last administration of the study drug and voluntarily adopt appropriate and effective contraceptive measures (non-oral contraceptives);
* Have a full understanding of this study, voluntarily participate in the trial, and voluntarily sign the written informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* Subjects with special dietary requirements who cannot adhere to a uniform diet;
* Subjects suspected or confirmed to be allergic to any component similar to the study drug or any ingredient in the study drug, or individuals with an allergic constitution;
* Subjects with past or present severe diseases/abnormalities (including but not limited to cardiac/cerebrovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatologic, malignant tumors, hematological, immunological, rheumatic, neurological or psychiatric diseases), or any acute or chronic disease or physiological condition that could interfere with the trial results;
* Subjects with severe infectious diseases within six months prior to screening, or a history of herpes zoster, disseminated herpes zoster, any infectious history judged by the investigator to likely worsen due to participation in the study, or any infectious history requiring antimicrobial treatment within two weeks after screening; or the presence of active infections, including acute and chronic infections as well as localized infections;
* Subjects with active or latent tuberculosis, or with a history of tuberculosis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | First dose of study drug up to 31 days after last dose of study drug
  Assessment by adverse event monitoring CTCAE 5.0

SECONDARY OUTCOMES:
Area Under the Curve（AUC） From Time Zero to Last Quantifiable Concentration | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72 hours following single dose administration;
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUC)last
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Pre dose and at 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, 72 hours following single dose administration;
  Time to Reach Maximum Observed Plasma Concentration (Tmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No